CLINICAL TRIAL: NCT05372354
Title: An Exploratory Phase 1b/2a Multicenter, Open-Label, Novel-Novel Combination Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of CC-92480 (BMS-986348) in Novel Therapeutic Combinations in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study to Evaluate Safety, Drug Levels and Effectiveness of CC-92480 (BMS-986348) in Combination With Other Treatments in Participants With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA057-003; 2023-509384-25 (Other: EU CTR); U1111-1269-5704 (Registry Identifier: WHO)
Record Dates: First submitted 2022-05-06; First posted 2022-05-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: BMS-986348; CC-92480; BMS-986158; Dexamethasone; Tazemetostat; Trametinib
MeSH Terms: conditions — Multiple Myeloma | interventions — tazemetostat; trametinib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 Arm A: Dose Finding (Experimental)
  Interventions: Drug: CC-92480; Drug: Tazemetostat; Drug: Dexamethasone
- Part 1 Arm B: Dose Finding (Experimental)
  Interventions: Drug: CC-92480; Drug: BMS-986158; Drug: Dexamethasone
- Part 1 Arm C: Dose Finding (Experimental)
  Interventions: Drug: CC-92480; Drug: Trametinib; Drug: Dexamethasone
- Part 2 Arm D: Dose Expansion (Active Comparator)
  Interventions: Drug: CC-92480; Drug: Dexamethasone
- Part 2 Arm E: Dose Expansion (Experimental)
  Interventions: Drug: CC-92480; Drug: Tazemetostat; Drug: Dexamethasone
- Part 2 Arm G: Dose Expansion (Experimental)
  Interventions: Drug: CC-92480; Drug: Trametinib; Drug: Dexamethasone

INTERVENTIONS:
Drug: CC-92480 — Specified dose on specified days
  Other Names: BMS-986348
Drug: Tazemetostat — Specified dose on specified days
  Arms: Part 1 Arm A: Dose Finding; Part 2 Arm E: Dose Expansion
Drug: BMS-986158 — Specified dose on specified days
  Arms: Part 1 Arm B: Dose Finding
Drug: Trametinib — Specified dose on specified days
  Arms: Part 1 Arm C: Dose Finding; Part 2 Arm G: Dose Expansion
Drug: Dexamethasone — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the safety, tolerability and preliminary effectiveness of CC-92480 (BMS-986348) in novel therapeutic combinations for the treatment of Relapsed or Refractory Multiple Myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory multiple myeloma (MM) and must:

  1. Have documented disease progression during or after their last myeloma therapy.
  2. For Part 1 Dose Finding: Be refractory to, intolerant to, or not a candidate for available, established therapies known to provide clinical benefit in MM; For Part 2 Dose Expansion: Be refractory to or have relapsed after the protocol specified number of prior lines of therapy that include an immunomodulatory drug (IMiD), a proteasome inhibitor, an anti-CD38 mAb, and a T-cell redirecting therapy (TRT, eg, a CAR-T or T-cell engaging bispecific treatment) unless the participant is not a candidate for TRT.
* Must have measurable disease.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
* Agree to follow the CC-92480 Pregnancy Prevention Plan (PPP).

Exclusion Criteria:

* Known active or history of central nervous system (CNS) involvement of MM
* Plasma cell leukemia; Waldenstrom's macroglobulinemia; polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes (POEMS) syndrome; or clinically significant light-chain amyloidosis.
* Impaired cardiac function or clinically significant cardiac disease
* Previous SARS-CoV-2 infection within 14 days for asymptomatic or mild symptomatic infections or 28 days for severe/critical illness prior to Cycle 1 Day 1 (C1D1)
* For Part 1: received prior therapy with CC-92480
* For Part 2: received prior therapy with CC-92480, tazemetostat, BMS-986158, or trametinib
* Previously received allogeneic stem-cell transplant at any time or received autologous stem-cell transplant within 12 weeks of initiating study treatment
* Received any of the following within 14 days prior to initiating study treatment:

  1. Plasmapheresis
  2. Major surgery
  3. Radiation therapy other than local therapy for myeloma associated bone lesions
  4. Use of any systemic anti-myeloma drug therapy
* Used any investigational agents within 28 days or 5 half-lives (whichever is shorter) prior to initiating study treatment
* COVID-19 vaccine within 14 days prior to C1D1

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2026-10-12 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From first participant first visit until 28 days after the last participant discontinues study treatment, up to approximately 4 years
Number of participants with Serious AEs | Up to approximately 4 years
Number of participants with AEs meeting protocol-defined DLT criteria | Up to approximately 4 years
Number of participants with AEs leading to discontinuation | Up to approximately 4 years
Number of deaths | Up to approximately 4 years
Establish recommended Phase 2 dose (RP2D) | Up to approximately 2 years
Establish dosing schedule of each combination for Part 2 Dose Expansion | Up to approximately 2 years

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 4 years
Very good partial response rate (VGPRR) | Up to approximately 4 years
Complete response rate (CRR) | Up to approximately 4 years
Time-to-response (TTR) | Up to approximately 4 years
Duration of response (DOR) | Up to approximately 4 years
Progression-free survival (PFS) | Up to approximately 4 years
Maximum observed plasma concentration (Cmax) | Up to approximately 28 days
Time to maximum plasma concentration (Tmax) | Up to approximately 28 days
Area under the concentration-time curve (AUC) | Up to approximately 28 days
Terminal Half-Life (T-Half) | Up to approximately 28 days
Apparent total body clearance (CLT/F) | Up to approximately 28 days
Apparent volume of distribution (Vz/F) | Up to approximately 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (5):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Johns Hopkins Medicine - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Canada (3):
  - Alberta Health Services AHS - Foothills Medical Centre FMC, Calgary, Alberta
  - University of Alberta - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network UHN - Princess Margaret Hospital PMH, Toronto, Ontario
- Oslo University Hospital, Oslo, Outside US and Canada, Norway
- Spain (3):
  - ICO - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
- United Kingdom (5):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Local Institution - 0001, Leicester, Leicestershire
  - Local Institution - 0014, Liverpool, Merseyside
  - Churchill Hospital, Oxford, Oxfordshire
  - NIHR UCLH Clinical Research Facility, London

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05372354.html